CLINICAL TRIAL: NCT05599451
Title: A Randomized, Controlled, Open-label, 4 Parallel Arms Study to Demonstrate Reductions in Exposure to Selected Harmful and Potentially Harmful Constituents (HPHC) of Cigarette (CIG) Smoke in Healthy Smokers Switching to Different Versions of Tobacco Heating System (THS) Compared to Continuing CIG Smoking, for 5 Days in Confinement
Brief Title: Reduced Exposure to HPHC in Smokers Switching From Cigarettes to Different Versions of THS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P1-REXC-10
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-05

CONDITIONS: Smoking; Tobacco Smoking; Tobacco Use
Keywords: Exposure Response; Smoking; Tobacco Heating System; Heated Tobacco
MeSH Terms: conditions — Smoking; Tobacco Smoking; Tobacco Use | interventions — Tobacco Products

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, open-label, 4 parallel arms study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- THS Blade device (Active Comparator): Subjects randomized to this arm participated in 5 days of ad libitum use, in confinement, of the THS Blade device (using regular THS blade tobacco sticks) between 06:30 AM and 11:00 PM.
  Interventions: Other: THS Blade device
- THS Induction Mono device (Active Comparator): Subjects randomized to this arm participated in 5 days of ad libitum use, in confinement, of the THS Induction Mono device (using regular THS induction tobacco sticks) between 06:30 AM and 11:00 PM.
  Interventions: Other: THS Induction Mono device
- THS Induction Mid device (Active Comparator): Subjects randomized to this arm participated in 5 days of ad libitum use, in confinement, of the THS Induction Mid device (using regular THS induction tobacco sticks) between 06:30 AM and 11:00 PM.
  Interventions: Other: THS Induction Mid device
- Cigarette (Active Comparator): Subjects randomized to this arm participated in 5 days of ad libitum use, in confinement, of the subject's preferred brand of regular (non-mentholated) cigarette between 06:30 AM and 11:00 PM.
  (Every subject brought a sufficient number of unopened, single-brand packs of CIG for the entire confinement period.)
  Interventions: Other: CIG

INTERVENTIONS:
Other: THS Blade device — Tobacco Heating System (THS) device with Blade technology for Blade tobacco stick use
  Other Names: IQOS (THS blade device); HEETS (blade heated tobacco sticks)
  Arms: THS Blade device
Other: THS Induction Mono device — Tobacco Heating System (THS) device with Induction technology (combined Charger-Holder device for Induction tobacco stick use).
  Other Names: IQOS Iluma One (THS induction device); TEREA (induction heated tobacco sticks)
  Arms: THS Induction Mono device
Other: THS Induction Mid device — Tobacco Heating System (THS) device with Induction technology (device with Induction stick Holder for Induction tobacco stick use and separate Charger).
  Other Names: IQOS Iluma (THS induction device); TEREA (induction heated tobacco sticks)
  Arms: THS Induction Mid device
Other: CIG — Subject's preferred brand of commercially available regular (non-mentholated) cigarettes. (Cigarettes are not provided by the study sponsor.)
  Other Names: Cigarette (non-mentholated)
  Arms: Cigarette

SUMMARY:
This was a randomized, controlled, open-label, 4 parallel arm study with a stratified randomization by sex (a quota for each sex [females and males] of at least 40% overall).

This study aimed to demonstrate the reduction of Biomarkers of Exposure (BoExp) to selected Harmful and Potentially Harmful Constituents (HPHC) in smokers switching from cigarettes (CIG) to each of the Tobacco Heating System (THS) variants with different heating technology (Blade device, Induction Mono device, or Induction Mid device, respectively), compared with smokers who continued to smoke CIG.

DETAILED DESCRIPTION:
Study Title: Reduced Exposure to Harmful and Potentially Harmful Constituents (HPHC) in Smokers Switching From Cigarettes to Different Versions of the Tobacco Heating System (THS)

Who carried out the research? This research was sponsored and funded by Philip Morris Products S.A.

What public involvement there was in the study? Ninety-one healthy, currently smoking, adults participated in this study.

Where and when the study took place? The study was conducted at a clinical trial facility managed by a contract research organization in Belfast, Northern Ireland, from November 4th 2022 to February 4th 2023.

Who participated in the study? Ninety-one healthy male or female adults, aged between 21 and 65 years, participated in this study. All participants were currently smoking. The participants did not plan to quit using tobacco and/or nicotine products within the next 3 months and had smoked continuously for at least the last 3 years prior to joining the study.

Each participant was given full and adequate oral and written information about the nature, purpose, possible risks, and benefits of the study. All participants received information on the risks of smoking, smoking cessation advice and a briefing on the Tobacco Heating System, for example, that its use is not risk-free.

Once each participant had received all the necessary information, and if they agreed to participate, this was documented in an Informed Consent Form with the date, time, and signature of both the participant and the study doctor. Participants were informed that they were free to withdraw from the study at any time.

What treatments or interventions did the participants take/receive? Eighty participants were randomly assigned to one of four study arms: THS Blade device, THS Induction Mono device, THS Induction Mid device, or Cigarette, for five days in a confinement setting.

Participants assigned to one of the THS arms or the Cigarette arm could use their assigned product, as often as they wished, from 6:30 AM to 11:00 PM during the five-day confinement period.

Urine was collected from each participant for analysis, for each 24 hours, from Day -1 (the start of the confinement period) to Day 5 (until discharge at the morning of Day 6).

Participants were also asked to evaluate their experience of using their assigned products, using a product experience questionnaire. The questionnaire assessed the perceived effects experienced by Cigarette smokers switching to the THS Blade device, THS Induction Mono device, or THS Induction Mid device compared to the experience of subjects continuing Cigarette smoking.

What happened during the study? A presentation of THS (without product use) was made to the participants during the Screening visit. All participants received information on the risks of smoking, smoking cessation advice, and a briefing that the use of THS is not risk-free. Eligible participants, fulfilling all criteria for participation, returned to the investigational site for confirmation of eligibility at the Admission visit (Day -2).

On Day -2 (Admission), after eligibility criteria had been verified, subjects had a product test of the THS Blade device and Induction Mono device (with use of up to three THS tobacco sticks per device). All eligible participants were then enrolled and participants willing to continue their participation in the study started their confinement period of seven days.

On Day -1, participants were randomly assigned to one of four arms: THS Blade device, THS Induction Mono device, THS Induction Mid device, or Cigarette. Participants were informed about their randomization arm by the study site staff on Day 1 prior to the start of product use.

The Exposure period in confinement began on Day 1 and consisted of 5 days of at will use of the assigned product in the THS and Cigarette arms. Use of any tobacco/nicotine containing product other than the assigned product was not allowed.

Daily 24-hour urine was collected from Day -1 to Day 5 for HPHC analysis. On Day 1, use of THS or Cigarette smoking in the respective arms was not supposed to start before the end of 24-hour urine collection of Day -1. The 24-hour urine collection period for Day 5 ended in the morning of Day 6 prior to Discharge.

On Day -1 and on Days 1 to 5, participants completed questionnaires to assess the perceived effects experienced after switching to THS, compared to the experience of participants who continued Cigarette smoking.

During the confinement period, adherence to investigational product arm allocation (exclusive use of the assigned THS devices with designated sticks, or Cigarette smoking, respectively) was ensured by strict distribution of the devices, and of each stick/cigarette upon demand of the subject to the study site staff.

Any participant who wanted to attempt to quit using any tobacco or nicotine-containing product at any time during the study (that is, to quit THS use or Cigarette smoking) was encouraged to do so and was to be referred to appropriate medical services. This decision would not affect the participant's financial compensation, and the participant was to be considered as remaining in the study.

The Exposure period to the assigned investigational product (THS or Cigarette) ended at 11:00 PM on Day 5, followed by Discharge on Day 6 after completion of all study procedures. Participants were allowed to smoke Cigarettes or use other tobacco or nicotine-containing products, at their discretion, only after discharge from the study.

After discharge at Day 6 or from the day of an early termination, subjects entered a 3-day Safety follow-up period during which any adverse reactions reported by the participants were collected. The follow-up of adverse reactions ongoing at discharge was conducted by the investigational site.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed the ICF and is able to understand the information provided in the ICF.
* Subject has been a smoker for ≥3 years prior to the screening visit (smoking cessation attempts during this period, if any, did not last > 6 months in total).
* Subject has continuously smoked on average ≥10 commercially available regular CIGs/day over the last 4 weeks. Smoking status will be verified based on a urinary cotinine test (cotinine ≥200 ng/mL).
* Subject is healthy as judged by the Investigator based on available assessments from the screening period (e.g., safety laboratory, spirometry, vital signs, physical examination, ECG, and medical history).
* Subject does not plan to quit smoking within the next three months.

Exclusion Criteria:

* As per the Investigator's judgment, the subject cannot participate in the study for any reason other than medical (e.g., psychological, social reason).
* Subject is legally incompetent, or physically or mentally incapable of giving consent (e.g., in emergency situations, under guardianship, prisoners).
* Subject has a clinically relevant disease which requires medication (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, urological, immunological, pulmonary, and cardiovascular disease) or any other medical condition (including safety laboratory), which as per the judgment of the Investigator would jeopardize the safety of the subject.
* Subject experienced within 30 days prior to screening/admission a body temperature >37.5°C or an acute illness (e.g., upper respiratory-tract infection, viral infection, etc.) or the subject has a confirmed or suspected active COVID-19 infection (based on the signs and symptoms observed at the time of assessment)
* As per the Investigator's judgment, the subject has medical conditions which do or will require a medical intervention (e.g., start of treatment, surgery, hospitalization) during the study participation, which may interfere with the study participation and/or study results.
* Subject has relevant history of, or current asthma condition or COPD condition, and/or clinically significant findings.
* Subject has donated blood or received whole blood or blood products within 3 months.
* BMI < 18.5 kg/m2 or ≥ 32.0 kg/m2.
* Positive serology test for HIV 1/2, HBV, or HCV.
* Subject has a positive alcohol breath test and/or has a history of alcohol disorder that could interfere with their participation in the study.
* The subject has a positive urine drug test.
* Subject or one of their family members is a current or former employee of the tobacco or e-cigarette industry.
* Subject or one of their family members is an employee of the investigational site or of any other parties involved in the study.
* Subject has participated in another clinical study within 3 months.
* Subject has been previously screened or enrolled in this study.
* Subject is pregnant (does not have negative pregnancy tests at screening and at admission) or is breastfeeding.
* For women of childbearing potential only: subject does not agree to use an acceptable method of effective contraception.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-02-04 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devinda Weeraratne, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled But Not Randomized: Subjects who were enrolled, but were not randomized to a study arm.
- Cigarette: Subjects randomized to this arm participated in 5 days of ad libitum use, in confinement, of the subject's preferred brand of regular (non-mentholated) cigarette between 06:30 AM and 11:00 PM.
  (Every subject brought a sufficient number of unopened, single-brand packs of CIG for the entire confinement period.)
  CIG: Subject's preferred brand of commercially available regular (non-mentholated) cigarettes. (Cigarettes are not provided by the study sponsor.)
Period: Overall Study
Arm/Group | Enrolled But Not Randomized | Cigarette | THS Blade Device | THS Induction Mono Device | THS Induction Mid Device
Started | 11 | 19 | 20 | 21 | 20
Completed | 0 | 19 | 20 | 20 | 20
Not Completed | 11 | 0 | 0 | 1 | 0
Not completed — Not randomized | 11 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cigarette | THS Blade Device | THS Induction Mono Device | THS Induction Mid Device | Total
Number analyzed (Participants) | 19 | 20 | 21 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (9.51) | 37.8 (10.96) | 40.0 (11.77) | 39.3 (9.19) | 38.8 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 12 | 11 | 43
  Male | 9 | 10 | 9 | 9 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18 | 20 | 21 | 20 | 79
  Black | 0 | 0 | 0 | 0 | 0
  Pacific Islander | 1 | 0 | 0 | 0 | 1
BMI (at screening) [Mean (Full Range); unit: kg/m²] | 26.19 [20.6 to 30.9] | 24.51 [19.6 to 30.7] | 25.35 [20.7 to 31.9] | 26.73 [21.7 to 30.5] | 25.69 [19.6 to 31.9]

OUTCOME MEASURES:

1. Primary Outcome: Concentration of 3-hydroxypropylmercapturic Acid (3-HPMA)
Description: Concentrations measured in urine, adjusted for creatinine, at Day 5. Geometric Least Squares means are provided for biomarkers of exposure (BoExp) in smokers switching from CIG to various THS versions (THS Blade device; THS Induction Mono device; THS Induction Mid device) compared to continuing CIG smoking for 5 days.
Time Frame: 5 days
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mg creatinine
Arm/Group | Cigarette | THS Blade Device | THS Induction Mono Device | THS Induction Mid Device
Number analyzed (Participants) | 19 | 20 | 21 | 20
ng/mg creatinine
  Baseline | 786.07 [605.60 to 1020.32] | 674.08 [478.57 to 949.46] | 781.63 [611.65 to 998.85] | 765.28 [579.16 to 1011.21]
  After 1 day | 711.21 [554.98 to 911.41] | 206.87 [163.28 to 262.09] | 223.71 [181.65 to 275.52] | 204.79 [164.80 to 254.48]
  After 2 days | 810.16 [589.94 to 1112.57] | 235.60 [185.92 to 298.56] | 235.20 [190.35 to 290.62] | 231.39 [187.62 to 285.39]
  After 3 days | 775.24 [558.75 to 1075.61] | 190.61 [146.36 to 248.24] | 199.11 [167.67 to 236.45] | 200.33 [158.43 to 253.31]
  After 4 days | 921.78 [715.95 to 1186.79] | 244.63 [195.86 to 305.53] | 231.94 [192.84 to 278.97] | 200.21 [153.50 to 261.12]
  After 5 days | 760.37 [581.14 to 994.87] | 227.64 [178.70 to 289.98] | 196.90 [155.34 to 249.56] | 211.03 [172.20 to 258.62]

2. Primary Outcome: Concentration of 2-cyanoethyl Mercapturic Acid N-acetyl-S-(2-cyanoethyl)-L-cysteine (2-CyEMA)
Description: as for outcome 1
Time Frame: 5 days
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mg creatinine
Arm/Group | Cigarette | THS Blade Device | THS Induction Mono Device | THS Induction Mid Device
Number analyzed (Participants) | 19 | 20 | 21 | 20
ng/mg creatinine
  Baseline | 96.01 [67.06 to 137.46] | 85.66 [57.14 to 128.42] | 107.33 [84.22 to 136.77] | 104.62 [79.50 to 137.68]
  After 1 day | 100.15 [76.73 to 130.71] | 27.81 [17.19 to 45.01] | 38.17 [30.22 to 48.22] | 32.93 [25.54 to 42.46]
  After 2 days | 106.01 [76.19 to 147.51] | 16.44 [10.40 to 25.96] | 21.38 [15.19 to 30.10] | 21.48 [16.90 to 27.30]
  After 3 days | 108.76 [78.01 to 151.63] | 13.31 [8.02 to 22.12] | 16.85 [11.93 to 23.81] | 18.09 [14.20 to 23.05]
  After 4 days | 113.99 [86.97 to 149.40] | 11.54 [7.19 to 18.53] | 13.74 [9.26 to 20.40] | 13.36 [9.75 to 18.31]
  After 5 days | 108.64 [81.43 to 144.96] | 12.20 [7.60 to 19.58] | 13.34 [8.80 to 20.22] | 15.95 [12.48 to 20.38]

3. Primary Outcome: Concentration of Monohydroxybutenyl Mercapturic Acid (MHBMA)
Description: as for outcome 1
Time Frame: 5 days
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mg creatinine
Arm/Group | Cigarette | THS Blade Device | THS Induction Mono Device | THS Induction Mid Device
Number analyzed (Participants) | 19 | 20 | 21 | 20
ng/mg creatinine
  Baseline | 2.08 [1.38 to 3.14] | 2.09 [1.39 to 3.12] | 1.37 [0.77 to 2.43] | 2.64 [1.92 to 3.63]
  After 1 day | 1.74 [1.21 to 2.52] | 0.43 [0.32 to 0.57] | 0.36 [0.24 to 0.55] | 0.52 [0.41 to 0.66]
  After 2 days | 2.19 [1.46 to 3.29] | 0.14 [0.11 to 0.18] | 0.15 [0.11 to 0.19] | 0.16 [0.13 to 0.20]
  After 3 days | 1.88 [1.20 to 2.93] | 0.08 [0.06 to 0.11] | 0.08 [0.06 to 0.10] | 0.10 [0.08 to 0.13]
  After 4 days | 2.01 [1.32 to 3.05] | 0.08 [0.06 to 0.10] | 0.09 [0.07 to 0.11] | 0.09 [0.07 to 0.11]
  After 5 days | 1.97 [1.34 to 2.91] | 0.10 [0.08 to 0.13] | 0.10 [0.08 to 0.12] | 0.10 [0.08 to 0.12]

4. Primary Outcome: Concentration of Total 4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol (Total NNAL)
Description: as for outcome 1
Time Frame: 5 days
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mg creatinine
Arm/Group | Cigarette | THS Blade Device | THS Induction Mono Device | THS Induction Mid Device
Number analyzed (Participants) | 19 | 20 | 21 | 20
pg/mg creatinine
  Baseline | 115.30 [83.91 to 158.43] | 101.92 [57.26 to 181.43] | 135.02 [96.24 to 189.43] | 150.11 [117.61 to 191.60]
  After 1 day | 104.20 [74.45 to 145.84] | 51.32 [28.62 to 92.05] | 82.04 [56.15 to 119.88] | 77.92 [58.24 to 104.24]
  After 2 days | 131.69 [89.40 to 194.00] | 42.43 [24.09 to 74.74] | 66.40 [43.62 to 101.10] | 68.00 [47.83 to 96.68]
  After 3 days | 127.57 [88.64 to 183.60] | 37.74 [20.39 to 69.85] | 63.40 [43.18 to 93.10] | 59.96 [43.31 to 83.02]
  After 4 days | 133.05 [94.47 to 187.38] | 34.49 [19.86 to 59.89] | 52.35 [35.97 to 76.20] | 54.24 [38.67 to 76.06]
  After 5 days | 127.04 [88.57 to 182.22] | 32.48 [17.70 to 59.61] | 53.63 [36.41 to 78.99] | 55.82 [40.88 to 76.22]

5. Primary Outcome: Levels of Carboxyhemoglobin (COHb)
Description: Carboxyhemoglobin (COHb) is assayed from whole blood. Expressed as % of saturation of hemoglobin. Blood measurements performed in the evening of Day 5. Geometric Least Squares means are provided for biomarkers of exposure (BoExp) in smokers switching from CIG to various THS versions (THS Blade device; THS Induction Mono device; THS Induction Mid device) compared to continuing CIG smoking for 5 days.
Time Frame: 5 days
Measure: Geometric Mean (95% Confidence Interval); unit: % in blood
Arm/Group | Cigarette | THS Blade Device | THS Induction Mono Device | THS Induction Mid Device
Number analyzed (Participants) | 19 | 20 | 21 | 20
% in blood
  Baseline | 5.26 [4.6 to 6.0] | 4.79 [4.0 to 5.8] | 5.17 [4.6 to 5.8] | 5.26 [4.6 to 6.0]
  After 1 day | 5.10 [4.5 to 5.8] | 1.50 [1.4 to 1.6] | 1.60 [1.3 to 1.9] | 1.60 [1.4 to 1.8]
  After 2 days | 5.29 [4.4 to 6.4] | 1.51 [1.3 to 1.7] | 1.59 [1.4 to 1.9] | 1.88 [1.5 to 2.4]
  After 3 days | 5.07 [4.3 to 5.9] | 1.33 [1.2 to 1.5] | 1.77 [1.4 to 2.2] | 1.84 [1.4 to 2.4]
  After 4 days | 4.77 [4.1 to 5.6] | 1.46 [1.3 to 1.7] | 1.66 [1.3 to 2.1] | 1.56 [1.4 to 1.7]
  After 5 days | 4.98 [4.1 to 6.0] | 1.38 [1.2 to 1.7] | 1.62 [1.3 to 2.0] | 1.78 [1.4 to 2.2]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signature of the ICF by each subject until the end of the safety follow-up period, a total duration for each subject of up to 39 days.
Arm/Group | Cigarette | THS Blade Device | THS Induction Mono Device | THS Induction Mid Device | Enrolled But Not Randomized
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20 | 0/21 | 0/20 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/21 | 0/20 | 0/11
Other Adverse Events (participants affected / at risk) | 0/19 | 9/20 | 1/21 | 5/20 | 0/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cigarette (N=19) | THS Blade Device (N=20) | THS Induction Mono Device (N=21) | THS Induction Mid Device (N=20) | Enrolled But Not Randomized (N=11)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Lip Dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT05599451/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/51/NCT05599451/SAP_001.pdf